CLINICAL TRIAL: NCT03804268
Title: A Phase 3, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of AGN-190584 in Participants With Presbyopia
Brief Title: Efficacy Study of Pilocarpine HCl Ophthalmic Solution (AGN-190584) in Participants With Presbyopia
Acronym: GEMINI 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1883-301-013
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle (Placebo Comparator): Participants received one drop of vehicle in each eye, once daily, for up to 30 days.
  Interventions: Other: Vehicle
- Pilocarpine HCl Ophthalmic Solution (Experimental): Participants received one drop of pilocarpine HCl ophthalmic solution 1.25% in each eye, once daily, for up to 30 days.
  Interventions: Drug: Pilocarpine HCl Ophthalmic Solution

INTERVENTIONS:
Other: Vehicle — Vehicle, one drop in each eye, once daily, for up to 30 days.
  Arms: Vehicle
Drug: Pilocarpine HCl Ophthalmic Solution — Pilocarpine HCl ophthalmic solution 1.25%, one drop in each eye, once daily, for up to 30 days.
  Other Names: AGN-190584; VUITY
  Arms: Pilocarpine HCl Ophthalmic Solution

SUMMARY:
A study to evaluate the efficacy, safety, and pharmacokinetics of pilocarpine hydrochloride (HCl) ophthalmic solution (AGN-190584) when administered bilaterally, once daily for 30 days in participants with presbyopia.

ELIGIBILITY:
Inclusion Criteria:

- Subjective complaints of poor near vision that impact activities of daily living

Exclusion Criteria:

* History of cataract surgery, phakic intraocular lens surgery, corneal inlay surgery, radial keratotomy, or any intraocular surgery
* Use of any topical ophthalmic medications, including artificial tears other than the study medications during the study
* Use of temporary or permanent punctal plugs or history of punctal cautery in one or both eyes
* Corneal abnormalities (including keratoconus, corneal scar, Fuchs' endothelial dystrophy, guttata, or edema) in either eye that are likely to interfere with visual acuity
* Narrow iridocorneal angles (Shaffer grade ≤2 or lower on gonioscopy examination), history of angle-closure glaucoma, or previous iridotomy
* Diagnosis of any type of glaucoma or ocular hypertension

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Safyan, Study Director — Allergan
Locations (36):
- United States (36):
  - Arizona Eye Center, Chandler, Arizona
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Assil Eye Institute, Beverly Hills, California
  - American Institute of Research, Los Angeles, California
  - Eye Research Foundation, Newport Beach, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Grutzmacher & Lewis, A Medical Corporation DBA Sacramento Eye Consultants, Sacramento, California
  - Haas Vision Center, Colorado Springs, Colorado
  - Danbury Eye Physicians and Surgeons P.C., Danbury, Connecticut
  - The Eye Associates, Bradenton, Florida
  - Bruce Segal, MD, Delray Beach, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - Florida Eye Associates, Melbourne, Florida
  - USF Eye Institute, Tampa, Florida
  - Price Vision Group, Indianapolis, Indiana
  - Sabates Eye Centers, Leawood, Kansas
  - The Eye Care Institute, Louisville, Kentucky
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Tauber Eye Center, Kansas City, Missouri
  - Alterman, Modi & Wolter, Poughkeepsie, New York
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Mundorf Eye Center, Charlotte, North Carolina
  - The Ohio State University, Columbus, Ohio
  - EyeCare Professionals DWA Insight Research Clinic, LLC, Powell, Ohio
  - Devers Eye Institute, Portland, Oregon
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Southern College of Optometry, Memphis, Tennessee
  - Nashville Vision Associates, Nashville, Tennessee
  - Hill Country Eye Center, Cedar Park, Texas
  - Key-Whitman Eye Center, Dallas, Texas
  - PNV Clinical Research LLC, San Antonio, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Hoopes, Durrie, Rivera Research, Draper, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lievens CW, Hom MM, McLaurin EB, Yuan J, Safyan E, Liu H. Pilocarpine HCl 1.25% for treatment of presbyopia after laser vision correction: pooled analysis of two phase 3 randomized trials (GEMINI 1 and 2). J Cataract Refract Surg. 2024 Jan 1;50(1):57-63. doi: 10.1097/j.jcrs.0000000000001313. PMID 37702453
- [Derived] Westheimer G. Topical Review: Pilocarpine-induced Miosis as Help for Early Presbyopes? Optom Vis Sci. 2022 Aug 1;99(8):632-634. doi: 10.1097/OPX.0000000000001924. Epub 2022 Jul 14. PMID 35848990
- [Derived] Waring GO 4th, Price FW Jr, Wirta D, McCabe C, Moshirfar M, Guo Q, Gore A, Liu H, Safyan E, Robinson MR. Safety and Efficacy of AGN-190584 in Individuals With Presbyopia: The GEMINI 1 Phase 3 Randomized Clinical Trial. JAMA Ophthalmol. 2022 Apr 1;140(4):363-371. doi: 10.1001/jamaophthalmol.2022.0059. PMID 35238902

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilocarpine HCl Ophthalmic Solution: Participants received one drop of pilocarpine hydrochloride (HCl) ophthalmic solution 1.25% in each eye, once daily, for up to 30 days.
Period: Overall Study
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Started | 160 | 163
Completed | 153 | 161
Not Completed | 7 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution | Total
Number analyzed (Participants) | 160 | 163 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (3.23) | 49.5 (3.81) | 49.6 (3.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 113 | 235
  Male | 38 | 50 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 31 | 57
  Not Hispanic or Latino | 134 | 132 | 266
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 13 | 25
  White | 144 | 148 | 292
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Gaining 3 Lines or More in Mesopic, High-contrast, Binocular Distance-Corrected Near Visual Acuity (DCNVA) at Day 30, Hour 3
Description: Visual acuity for near (40 centimeters (cm)) target was measured in mesopic conditions using an eye chart. Mesopic condition was defined as low lighting 3.2 to 3.5 candelas per square meter (cd/m^2) measured at the target. Percentage of participants with 3 lines or more improvement from Baseline in mesopic, high-contrast DCNVA are reported.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: Intent-to-treat (ITT) Population included all randomized participants. Missing data was imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 160 | 163
percentage of participants | 8.1 | 30.7
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p < 0.0001, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 22.5, 95% CI 2-sided [14.3 to 30.8] — Analysis was done using Chi-square test. 95% confidence interval for the percentage differences was calculated based on the normal approximation based on pooled variance without continuity correction

2. Secondary Outcome: Percentage of Participants Gaining 3 Lines or More in Mesopic, High-contrast, Binocular Distance-Corrected Near Visual Acuity (DCNVA) at Day 30, Hour 6
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions using an eye chart. Mesopic condition was defined as low lighting 3.2 to 3.5 candelas per square meter measured at the target. Percentage of participants with 3 lines or more improvement from Baseline in mesopic, high-contrast DCNVA are reported.
Time Frame: Baseline (Day 1) to Day 30 (Hour 6)
Population: ITT Population included all randomized participants. Missing data was imputed as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Pilocarpine HCl Ophthalmic Solution: Participants received one drop of pilocarpine HCl ophthalmic solution1.25% in each eye, once daily, for up to 30 days.
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 160 | 163
percentage of participants | 8.8 | 18.4
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 9.7, 95% CI 2-sided [2.3 to 17.0] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Gaining 3-lines or More in Mesopic, High-contrast, Binocular, DCNVA at Day 30, Hour 8
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Day 30 (Hour 8)
Population: ITT Population included all randomized participants. Overall number analyzed is the number of participants with data available for analyses at Baseline and the timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 153 | 161
percentage of participants | 8.5 | 10.6
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 1.0000, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 2.1, 95% CI 2-sided [-4.4 to 8.5] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Mesopic, High-contrast, Binocular DCNVA Letters at Day 30, Hour 0.5
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions using an eye chart. Mesopic condition was defined as low lighting 3.2 to 3.5 cd/m^2 measured at the target. A positive change from Baseline indicates improvement in visual acuity. Mixed effect model for repeated measures (MMRM) was used for analyses.
Time Frame: Baseline (Day 1) to Day 30 (Hour 0.5)
Population: ITT Population included all randomized participants. Overall number analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: letters read correctly
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 153 | 158
letters read correctly | 4.2 (0.55) | 9.3 (0.54)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, MMRM — MMRM with fixed effects: study intervention group,visit,visit by study intervention group interaction,age group,Baseline binocular DCNVA severity,iris color,emmetrope/non-emmetrope, Baseline value, and Baseline value by visit interaction was used; P-value was adjusted for multiplicity control; Least Square (LS) Mean Difference = 5.1, 95% CI 2-sided [3.7 to 6.5], Standard Error of Mean 0.72

5. Secondary Outcome: Percentage of Participants Achieving 20/40 or Better in Photopic, High-contrast, Binocular, DCNVA at Day 30, Hour 1
Description: Visual acuity for near (40 cm) target was measured in photopic conditions using an eye chart. Photopic condition was defined as high lighting ≥80 cd/m^2 measured at the target. Percentage of participants achieving 20/40 or better in photopic, high-contrast, binocular, DCNVA are reported.
Time Frame: Day 30 (Hour 1)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 153 | 161
percentage of participants | 73.9 | 92.5
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 18.7, 95% CI 2-sided [10.6 to 26.7] — Analysis was done using Chi-square test. 95% confidence interval was calculated based on normal approximation based on pooled variance without continuity correction

6. Secondary Outcome: Mean Change From Baseline in Mesopic Near Vision Presbyopia Task-based Questionnaire (NVPTQ) Performance Score at Day 30, Hour 3
Description: NVPTQ had 12 questions on 4 reading tasks(reading a paragraph from book, excerpts from an article in newspaper, portion of a nutrition label, and a section from restaurant menu). Participants completed specific reading tasks under mesopic conditions without any near-vision correction and answered 3 questions for each task, rating their vision-related reading ability as 0=I could not read any text due to problems seeing up close,1=poor,2=fair,3=good,4=very good,5=excellent;impact of squinting on performance as 0=No,I did not squint, 1=Yes,squinting helped me read some/all text, 2=Yes,but I still could not read any of the text; and satisfaction as 0=very dissatisfied to 4=very satisfied. The score based on vision related ability and impact of squinting=(Book testlet+Newspaper testlet+Menu testlet+Nutrition Label testlet)/(testlets with non-missing responses), total possible score of 0-5. Higher scores=better outcomes;positive change from Baseline=improved performance(reading ability).
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: ITT Population included all randomized participants. Overall number analyzed is the number of participants with data available for analyses. Analysis of Covariance (ANCOVA) was used for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 148 | 154
score on a scale | 0.6 (0.11) | 1.4 (0.11)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, ANCOVA — Analysis of covariance (ANCOVA) was used with study intervention group, age group, Baseline binocular DCNVA severity, iris color (brown/non-brown), emmetrope/non-emmetrope, and Baseline domain score as fixed effects; P-value was adjusted for multiplicity control; LS Mean Difference = 0.8, 95% CI 2-sided [0.6 to 1.1], Standard Error of Mean 0.14

7. Secondary Outcome: Change From Baseline in Photopic, High-contrast, Binocular Distance-corrected Intermediate Visual Acuity (DCIVA) Letters at Day 30, Hour 3
Description: Visual acuity for intermediate (66 cm) target was measured in photopic conditions using an eye chart. Photopic condition was defined as high lighting ≥80 cd/m^2 measured at the target. A positive change from Baseline indicates improvement in visual acuity. MMRM was used for analyses.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: letters read correctly
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 153 | 161
letters read correctly | 3.1 (0.42) | 6.6 (0.41)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, MMRM — [p-value comment as in outcome 4, analysis 1]; P-value was adjusted for multiplicity control; LS Mean Difference = 3.5, 95% CI 2-sided [2.4 to 4.6], Standard Error of Mean 0.55

8. Secondary Outcome: Percentage of Participants Gaining 3-lines or More in Mesopic, High-contrast, Binocular, DCNVA at Day 30, Hour 10
Description: Visual acuity for near (40cm) target was measured in mesopic conditions using an eye chart. Mesopic condition was defined as low lighting 3.2 to 3.5 cd/m^2measured at the target. Percentage of participants with 3 lines or more improvement from Baseline in mesopic, high-contrast, binocular DCNVA are reported.
Time Frame: Baseline (Day1) to Day 30 (Hour 10)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 152 | 160
percentage of participants | 8.6 | 7.5
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 1.0000, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = -1.1, 95% CI 2-sided [-7.1 to 5.0] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in Mesopic, High-contrast, Binocular DCNVA Letters at Day 30, Hour 0.25
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions. Mesopic condition was defined as low lighting 3.2 to 3.5 cd/m^2 measured at the target. A positive change from Baseline indicates improvement in visual acuity. MMRM was used for analyses.
Time Frame: Baseline (Day 1) to Day 30 (Hour 0.25)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: letters correctly read
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 153 | 158
letters correctly read | 3.7 (0.50) | 6.3 (0.49)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, MMRM — [p-value comment as in outcome 4, analysis 1]; P-value was adjusted for multiplicity control; LS Mean Difference = 2.6, 95% CI 2-sided [1.3 to 3.9], Standard Error of Mean 0.66

10. Secondary Outcome: Percentage of Participants Achieving 20/40 or Better in Photopic, High-contrast, Binocular, DCNVA at Day 30, Hour 3
Description: Visual acuity for near (40 cm) target was measured in mesopic conditions using an eye chart. Photopic condition was defined as high lighting ≥80 cd/m^2 measured at the target. Percentage of participants achieving 20/40 or better in photopic, high-contrast, binocular, DCNVA are reported.
Time Frame: Day 30 (Hour 3)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 153 | 161
percentage of participants | 71.9 | 84.5
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0171, Chi-squared — P-value was adjusted for multiplicity control; Percentage Difference = 12.6, 95% CI 2-sided [3.5 to 21.6] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Mean Change From Baseline in Mesopic NVPTQ Satisfaction Score at Day 30, Hour 3
Description: NVPTQ had 12 questions on 4 reading tasks(reading a paragraph from book, excerpts from an article in newspaper, portion of a nutrition label, and a section from restaurant menu). Participants completed specific reading tasks under mesopic conditions without any near-vision correction and answered 3 questions for each task, rating their vision-related reading ability as 0=I could not read any text due to problems seeing up close to 5=excellent; impact of squinting on performance as 0=No, I did not squint, 1=Yes, squinting helped me read some/all text, 2=Yes, but I still could not read any of the text; and satisfaction as 0=very dissatisfied,1=dissatisfied,2=neither satisfied nor dissatisfied,3=satisfied, 4=very satisfied. The score based on satisfaction items=(Book testlet+Newspaper testlet+Menu testlet+Nutrition Label testlet)/(testlets with non-missing responses) for a total possible score of 0 to 4. Higher scores=better outcomes; a positive change from Baseline=higher satisfaction.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: ITT Population included all randomized participants. Overall number analyzed is the number of participants with data available for analyses. ANCOVA was used for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 148 | 154
score on a scale | 0.6 (0.11) | 1.4 (0.10)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, ANCOVA — ANCOVA was used with study intervention group, age group, baseline binocular DCNVA severity, iris color (brown/non-brown), emmetrope/non-emmetrope, and baseline domain score as fixed effects; P-value was adjusted for multiplicity control; LS Mean Difference = 0.8, 95% CI 2-sided [0.5 to 1.1], Standard Error of Mean 0.13

12. Secondary Outcome: Mean Change From Baseline in Presbyopia Impact and Coping Questionnaire (PICQ) Coping Score at Day 30, Hour 3
Description: PICQ=20 questions about impact experienced by participants due to their problems over past 7 days.PICQ Coping domain had 8 items: 1:Normal-sized text,2:Small-sized text,3:Information on a computer,4:Information on a cell phone,5:Increase font size,6:Use glasses to read close,12:Hold reading materials farther out/closer,13:Squint to read. Each item had response categories:0=never to 4=all the time. Items 3, 4, 5, and 6 had additional response categories with values of 9/10 to indicate the question is not applicable to participant and were assigned missing values.PICQ Coping Score:(Item 1,2 Testlet+Item 3,4 Testlet+Item 5+Item 6+Item 12+Item 13)/non-missing responses to the 6 components of coping score where Items 1,2 Testlet=(Item1+Item2)/non-missing responses to Items 1,2;Items 3,4 Testlet=(Item3+Item4)/non-missing responses to Items 3, 4. Score ranges:0=to least amount of coping to 4=greatest amount of coping. Higher scores=poorer outcome; a negative change from Baseline=improvement.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 148 | 159
score on a scale | -0.5 (0.07) | -1.0 (0.07)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value was adjusted for multiplicity control; LS Mean Difference = -0.5, 95% CI 2-sided [-0.6 to -0.3], Standard Error of Mean 0.09

13. Secondary Outcome: Mean Change From Baseline in PICQ Impact Score at Day 30, Hour 3
Description: PICQ had 20 questions about impact experienced by participants due to their problems seeing up over past 7 days. PICQ Impact domain had 6 items: Item 9:Rely on others,15:rest eyes,16:Feel older,17:Feel self-conscious,19:Take longer to complete a task,20:Inconvenient. First 5 impacts items included response categories: 0=never to 4=all the time. Item 20 had response categories: 0=not at all to 4=extremely. Item 9 included an additional response category with a value of 9 to indicate question was not applicable to participant and the responses were assigned missing values. PICQ Impacts Score=[(Item9+Item15+Items16,17Testlet+Item19+Item20)/(nonmissing responses to 5 components of impacts score)] where Items 16,17 Testlet=(Item16+Item17)/non-missing responses to Items 16 and 17. PICQ Impact score ranges from 0 to 4; with 0=least amount of impacts to 4=greatest amount of impacts. Higher scores correspond to poorer outcomes. A negative change from Baseline=improvement.
Time Frame: Baseline (Day 1) to Day 30 (Hour 3)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
Number analyzed (Participants) | 148 | 159
score on a scale | -0.4 (0.06) | -0.7 (0.06)
Statistical Analysis 1: Comparison: Vehicle vs Pilocarpine HCl Ophthalmic Solution; Test type: Superiority; p = 0.0114, ANCOVA — [p-value comment as in outcome 11, analysis 1]; P-value was adjusted for multiplicity control; LS Mean Difference = -0.3, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.08

ADVERSE EVENTS:
Time Frame: First dose of study drug intervention to within 30 days after last dose (Up to 60 days)
Description: All-cause Mortality: All enrolled participants. Serious Adverse Events and Other (non-serious) Adverse Events: Safety Population included all participants who received at least 1 administration of study intervention.
Arm/Group | Vehicle | Pilocarpine HCl Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/163
Other Adverse Events (participants affected / at risk) | 15/159 | 23/163
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=159) | Pilocarpine HCl Ophthalmic Solution (N=163)
Headache (Nervous system disorders) | 15 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT03804268/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT03804268/SAP_001.pdf